CLINICAL TRIAL: NCT03295474
Title: Telemonitoring in Pulmonary Rehabilitation: Feasibility and Acceptability of a Remote Pulse Oxymetry System (FA-TELE-REHAB)
Brief Title: Telemonitoring in Pulmonary Rehabilitation: Feasibility and Acceptability of a Remote Pulse Oxymetry System.
Status: Completed | Type: Observational
Sponsor: ADIR Association (Other)
Responsible Party: Sponsor
Other Study IDs: FA-TELE-REHAB
Record Dates: First submitted 2017-09-25; First posted 2017-09-27 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-01

CONDITIONS: Chronic Obstructive Pulmonary Disease; Pulmonary Rehabilitation; Telemedicine
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rehabilitation using telehealth technology
  Interventions: Other: Rehabilitation using telehealth technology

INTERVENTIONS:
Other: Rehabilitation using telehealth technology — Consecutive patients with chronic respiratory disease referred for pulmonary rehabilitation are offered to participate in the protocol.
  Patients are taught to use the system during the first session of aerobic training.
  During 2 to 5 sessions of aerobic training (depending on the number of sessions needed to be autonomous), they are monitored in the pulmonary rehabilitation center with an oximeter device (Nonin 3150).
  At the end of every session, patients are asked to answer to 3 questions on a Likert scale (see outcome session).
  The therapist also ascertains wether the telemonitoring gateway successfully provided informations regarding the session.
  The study takes off on the session during which the patients are autonomous in using the telehealthcare system.
  If patients are not autonomous on the fifth session, the study also takes off.

SUMMARY:
Pulmonary rehabilitation effectively improves outcomes in patients with chronic respiratory disease, however there is a lack of pulmonary rehabilitation centers. Telehealth technology is one solution to deliver supervised home-based rehabilitation (tele-rehabilitation).

However, the feasibility and the acceptability of using telehealth technology to deliver tele-rehabilitation has not been assessed in a large scale multicenter study.

Therefore, the aim of this study is to assess the feasibility and the acceptability of telemonitoring system during pulmonary rehabilitation in patients with chronic respiratory disease.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years ;
* Referred for pulmonary rehabilitation (every chronic respiratory disease accepted).

Exclusion Criteria:

* Pregnant woman or likely to be ;
* Patient under guardianship ;
* Neuropathic disorder ;
* Contraindication to cardiopulmonary exercise testing or pulmonary rehabilitation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every patients referred for pulmonary rehabilitation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Ability of the patients to be autonomous when using the device. | 2 to 5 sessions for 100 different patients will be assessed for a total time frame a 1 year. Data will be collected after every sessions and presented as the number of patients autonomous when using the device
  Number of patients autonomous when using the device will be presented for the the 2nd, 3rd, 4th and 5th session.
Patient's satisfaction assessed by Likert scale. | 2 to 5 sessions for 100 different patients will be assessed for a total time frame a 1 year. Outcome will be assessed during the sessions of every patient
  Data will be presented as the patient's satisfaction of the system at the end of the 5 sessions
Reliability of the telemedicine gateway in providing data. | 2 to 5 sessions will be carried out for 100 patients for a total time frame of 1 year. For every patient, sessions will be carried out on separate days (with a minimum of 1 day of rest between sessions)
  Data will be collected at the end of every sessions. Final endpoint will be the reliability of the telemedicine Gateway in providing data through study completion.
  Calculation : number of sessions provided by telemedicine gateway/number of scheduled sessions

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Tardif, MD, Principal Investigator — CHU-Hôpitaux de Rouen - Hôpital de Bois-Guillaume, Service de physiologie urinaire, digestive, respiratoire et sportive, Bois-Guillaume, France; Cuvelier Antoine, Prof, PhD, Study Chair — CHU-Hôpitaux de Rouen - Service de pneumologie, Hôpital de Bois-Guillaume, Rouen, France ; UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France.; Tristan Bonnevie, MsC, Study Chair — ADIR Association, Bois-Guillaume, France ; UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France; Francis-Edouard Gravier, PT, Study Chair — ADIR Association, Bois-Guillaume, France; Catherine Viacroze, MD, Study Chair — CHU-Hôpitaux de Rouen - Hôpital de Bois-Guillaume, Service de pneumologie, Bois-Guillaume, France; David Debeaumont, MD, Study Chair — CHU-Hôpitaux de Rouen - Hôpital de Bois-Guillaume, Service de physiologie urinaire, digestive, respiratoire et sportive, Bois-Guillaume, France; Jean-François Muir, Prof, PhD, Study Chair — CHU-Hôpitaux de Rouen - Service de pneumologie, Hôpital de Bois-Guillaume, Rouen, France ; UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France ; ADIR Association, Bois-Guillaume, France; Bouchra Lamia, Prof, PhD, Study Chair — UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France ; Service de pneumologie, Hôpital Jacques Monod 76290 Montivilliers; Jean Quieffin, MD, Study Chair — Service de pneumologie, Hôpital Jacques Monod 76290 Montivilliers; Guillaume Prieur, MsC, Study Chair — Service de pneumologie, Hôpital Jacques Monod 76290 Montivilliers.; Clément Médrinal, MsC, Study Chair — UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France. Service de réanimation, Groupe Hospitalier du Havre, France
Locations (2):
- France (2):
  - ADIR Association, Bois-Guillaume
  - Groupe Hospitalier du Havre, Le Havre

REFERENCES:
- [Derived] Bonnevie T, Gravier FE, Elkins M, Dupuis J, Prieur G, Combret Y, Viacroze C, Debeaumont D, Robleda-Quesada A, Quieffin J, Lamia B, Patout M, Cuvelier A, Muir JF, Medrinal C, Tardif C. People undertaking pulmonary rehabilitation are willing and able to provide accurate data via a remote pulse oximetry system: a multicentre observational study. J Physiother. 2019 Jan;65(1):28-36. doi: 10.1016/j.jphys.2018.11.002. Epub 2018 Dec 17. PMID 30573441